CLINICAL TRIAL: NCT07176767
Title: The IPAD Cohort Study: Insomnia and Positive Airway Pressure Adherence in Children and Adolescents
Acronym: IPAD
Status: Recruiting | Type: Observational
Sponsor: Lena Xiao (Other)
Collaborators: American Academy of Sleep Medicine (Other); The Hospital for Sick Children (SickKids) (Unknown)
Responsible Party: Sponsor-Investigator, Lena Xiao, Clinical Assistant Professor, University of British Columbia
Organization: University of British Columbia (Other)
Other Study IDs: H25-00289; 354-FP-24 (Other Grant/Funding Number: American Academy of Sleep Medicine Foundation)
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Sleep Apnea, Obstructive; Insomnia
Keywords: Obstructive Sleep Apnea; Insomnia; Pediatric Sleep; Positive Airway Pressure Adherence
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- OSA Children Starting PAP: Children aged 8-18 years old diagnosed with obstructive sleep apnea (OSA) who are to be initiated on Positive Airway Pressure (PAP) therapy. Children and their caregivers must be willing and able to complete questionnaires about sleep as well as physical and mental health.
  Interventions: Device: Positive airway pressure therapy

INTERVENTIONS:
Device: Positive airway pressure therapy — Initiation of continuous or bilevel positive airway pressure therapy
  Other Names: Continuous positive airway pressure therapy; Bilevel positive airway pressure therapy

SUMMARY:
Positive Airway Pressure (PAP) is a treatment used to help people with sleep-disordered breathing, particularly those with obstructive sleep apnea (OSA). The device delivers pressurized air through a mask to keep the airways open during sleep, improving breathing and preventing interruptions in sleep.

Studying how insomnia affects PAP adherence in children can help improve future treatments.

However, no long-term studies have looked at this in children. Based on previous research, the investigators plan to conduct a study across multiple centers focusing on children with OSA starting PAP therapy. The study will explore how insomnia affects PAP adherence and how race and ethnicity play a role.

DETAILED DESCRIPTION:
The first line of treatment for obstructive sleep apnea (OSA) is positive airway pressure (PAP) therapy, yet children have a less than 50% adherence rate, leaving many undertreated for this condition. Insomnia has been established as a modifiable risk factor for lowering PAP therapy adherence in adults with comorbid insomnia and sleep apnea (COMISA), and research has shown that treating insomnia with cognitive behavioural therapy for insomnia (CBTi) improved PAP adherence in adults. This is an important step forward for improving COMISA treatment outcomes, but cannot yet be applied to children without researching this relationship in paediatric populations. This study will address this research gap by conducting a thorough, in-depth evaluation of the association between paediatric COMISA and PAP adherence. The investigators aim to find whether a causal relationship exists between insomnia and PAP adherence in children with OSA, which has never been assessed longitudinally in children.

This multicenter study will be conducted at two tertiary care academic hospitals: The Hospital for Sick Children (Toronto, Canada) and British Columbia Children's Hospital (BCCH) (Vancouver, Canada). This study will include 82 participants from a diverse population to assess the association between race and ethnicity with PAP therapy adherence, based on previous research showing that being part of a self-identified minority is associated with lower PAP therapy adherence. Participants and caregivers will be asked to complete questionnaires regarding insomnia, sleep behaviour and quality of life at baseline prior to PAP therapy initiation. Electronic follow up questionnaires will be administered at 1, 2, and 3 months after PAP therapy initiation and PAP download data will be completed remotely. The primary objective of this study is to evaluate the impact of baseline insomnia on PAP therapy adherence at 3 months based on self-identified racial and ethnic minority. The results of this study will provide treatment insight and improvement to children with COMISA being treated with PAP therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 8-18 years old
2. Obstructive apnea-hypopnea index ≥ 5/hour on baseline diagnostic polysomnogram (PSG)
3. Newly prescribed PAP therapy

Exclusion Criteria:

1) Developmental disability precluding ability to answer questionnaires

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will be recruited from two tertiary care academic hospitals, The Hospital for Sick Children (Toronto, Canada) and British Columbia Children's Hospital (BCCH) (Vancouver, Canada).
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean minutes of nightly PAP usage | 90 days
  Adherence will be determined objectively using ventilator download data (days 60-90 after PAP initiation)

SECONDARY OUTCOMES:
Mean minutes of nightly PAP usage | 30, 60 days
  Adherence will be determined objectively using ventilator download data (days 0-30 and 30-60 after PAP initiation)
Self-Reported Sense of Mastery (Caregiver) | 0, 90 days
  The self-reported Pearlin Mastery Scale will be used to measure the caregiver's mastery. Scores range from 7 to 28, with higher scores indicating greater levels of mastery.
Self-Reported Sense of Mastery (Participant) | 0, 90 days
  The self-reported Pearlin Mastery Scale will be used to measure the participant's individual mastery. Scores range from 7 to 28, with higher scores indicating greater levels of mastery.
Self-Reported Psychological Scale (Percentage Rank) | 0, 90 days
  The self-reported Psychological Scale from the KIDSCREEN-10 questionnaire will be used to measure health-related quality of life. The score ranges from 10-50, with lower scores indicating a "dissatisfaction with life".
Self-Reported Psychological Scale | 0, 90 days
  The self-reported Psychological Scale from the Strengths and Difficulties questionnaire will be used. Scores range from 0-50 with higher scores indicating more difficulties and lower scores indicating more strengths.
Self-Reported Sleep Diary | 0, 90 days
  The self-reported National Institutes of Health (NIH) 1-week Sleep Diary will be used to record the quality and quantity of sleep.
Caregiver-Reported Insomnia Questionnaire | 0, 90 days
  The caregiver-reported Pediatric Insomnia Severity Index will be used to measure the severity of pediatric insomnia symptoms. Scores range from 0 to 30, with higher scores indicating greater insomnia severity.
Self-Reported Insomnia Questionnaire (Participant) | 0, 30, 60, 90 days
  The self-reported Insomnia Severity Index will be used to measure the nature, severity and impact of the participant's insomnia. Scores range from 0 to 28, with higher scores indicating greater insomnia severity.
Self-Reported Insomnia Questionnaire (Participant) | 0, 30, 60, 90 days
  The self-reported Insomnia Severity Index will be used to diagnose insomnia in the participant. Children will be classified as having insomnia using a cut-off of ≥ 9 points, based on the Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition.
Self-Reported Insomnia Questionnaire (Caregiver) | 0, 90 days
  The self-reported Insomnia Severity Index will be used to measure the nature, severity and impact of the caregiver's insomnia. Scores range from 0 to 28, with higher scores indicating greater insomnia severity.
Self-Reported Insomnia Questionnaire (Caregiver) | 0, 90 days
  The self-reported Insomnia Severity Index will be used to diagnose insomnia in the caregiver. Caregiver's will be classified as having insomnia using a cut-off of ≥ 9 points, based on the Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition.
Self-Reported Chronotype Questionnaire | 0, 90 days
  The self-reported Munich Chronotype Questionnaire will be used to measure participant chronotype. Scores range from 16 to 86 with scores below 42 indicating "evening types", scores between 42-58 indicating "intermediate types" and scores above 58 indicating "morning types".
Self-Reported Chronotype Questionnaire | 0, 90 days
  The self-reported Morningness/Eveningness Questionnaire will be used to measure differences in activeness and alertness in the mornings and evenings. Scores range from 16 to 86, with lower scores representing evening preference and higher scores representing morning preference.
Caregiver's Self-Reported Chronotype Questionnaire | 0, 90 days
  The self-reported Morningness/Eveningness Questionnaire will be used to measure the caregiver's differences in activeness and alertness in the mornings and evenings. Scores range from 16 to 86, with lower scores representing evening preference and higher scores representing morning preference.
Self-Reported Daytime Sleepiness Questionnaire | 0, 90 days
  The self-reported Epworth Sleepiness Scale will be used to measure daytime sleepiness. Scores range from 0-24 with lower score indicating less daytime sleepiness.
Self-Reported Caffeine Intake Questionnaire | 0, 90 days
  The self-reported Caffeine Consumption Questionnaire-Revised will be used to measure weekly caffeine intake. The quantity and frequency of caffeinated products reported is used to estimate the average daily caffeine consumption in mg.
Self-Reported Sleep Hygiene Questionnaire | 0, 90 days
  The self-reported Adolescent Sleep Hygiene Scale (ASHS) will be used to assess sleep habits and hygiene practices. The 33-item scale contains 28 quantitative items, which are scored as the following: never (0%) = 1; once in a while (20%) = 2; sometimes (40%) = 3; quite often (60%) = 4; frequently, if not always (80%) = 5; always (100%) = 6. Total scores range from 28-168, with higher scores indicating greater sleep hygiene.
Caregiver-Reported Global Rating Scale of Change | 90 days
  The caregiver-reported Global Rating Scale of Change will be used to measure the caregiver's perceived improvement or deterioration of the child's quality of life over time. The scale ranges from -7 to +7, with greater scores indicating improvements in quality of life.
Self-Reported Global Rating Scale of Change | 90 days
  The self-reported Global Rating Scale of Change will be used to measure the participant's perceived improvement or deterioration of their quality of life over time. The scale ranges from -7 to +7, with greater scores indicating improvements in quality of life.
Self-Reported PAP Adherence Questionnaire | 90 days
  The self-reported Adherence Barriers to CPAP Questionnaire will be used to estimate the participant's success or failure to use their PAP. The score ranges from 31 to 155, with greater scores indicating a higher number and severity of CPAP barriers.
Self-Reported Psychological (Total Anxiety) Subscale | 0, 90 days
  The self-reported Total Anxiety Subscale (major outcome) from the Revised Child Anxiety and Depression Scale will be used. The raw score from the subscale, which ranges from 0-45, will be used to calculate the T score by taking into consideration development level and gender. A T score of 65 or higher indicates a score borderline the clinical threshold and a T score of 70 or higher indicates a score above the clinical threshold.
Self-Reported Psychological (Total Depression) Scale | 0, 90 days
  The self-reported Total Depression (major outcome) from the Revised Child Anxiety and Depression Scale will be used. The raw score from the subscale, which ranges from 0-30, will be used to calculate the T score by taking into consideration development level and gender. A T score of 65 or higher indicates a score borderline the clinical threshold and a T score of 70 or higher indicates a score above the clinical threshold.
Self-Reported Psychological (Social Phobia) Scale | 0, 90 days
  The self-reported Social Phobia Subscale (major outcome) from the Revised Child Anxiety and Depression Scale will be used. The raw score from the subscale, which ranges from 0-27, will be used to calculate the T score by taking into consideration development level and gender. A T score of 65 or higher indicates a score borderline the clinical threshold and a T score of 70 or higher indicates a score above the clinical threshold.
Self-Reported Psychological (Panic Disorder) Scale | 0, 90 days
  The self-reported Panic Disorder Subscale (major outcome) from the Revised Child Anxiety and Depression Scale will be used. The raw score from the subscale, which ranges from 0-27, will be used to calculate the T score by taking into consideration development level and gender. A T score of 65 or higher indicates a score borderline the clinical threshold and a T score of 70 or higher indicates a score above the clinical threshold.
Self-Reported Psychological (Major Depression) Scale | 0, 90 days
  The self-reported Major Depression Subscale (major outcome) from the Revised Child Anxiety and Depression Scale will be used. The raw score from the subscale, which ranges from 0-30, will be used to calculate the T score by taking into consideration development level and gender. A T score of 65 or higher indicates a score borderline the clinical threshold and a T score of 70 or higher indicates a score above the clinical threshold.
Self-Reported Psychological (Separation Anxiety) Scale | 0, 90 days
  The self-reported Separation Anxiety Subscale (major outcome) from the Revised Child Anxiety and Depression Scale will be used. The raw score from the subscale, which ranges from 0-21, will be used to calculate the T score by taking into consideration development level and gender. A T score of 65 or higher indicates a score borderline the clinical threshold and a T score of 70 or higher indicates a score above the clinical threshold.
Self-Reported Psychological (Generalized Anxiety) Scale | 0, 90 days
  The self-reported Generalized Anxiety Subscale (major outcome) from the Revised Child Anxiety and Depression Scale will be used. The raw score from the subscale, which ranges from 0-18, will be used to calculate the T score by taking into consideration development level and gender. A T score of 65 or higher indicates a score borderline the clinical threshold and a T score of 70 or higher indicates a score above the clinical threshold.
Self-Reported Psychological (Obsessive-Compulsive) Scale | 0, 90 days
  The self-reported Obsessive-Compulsive Subscale (major outcome) from the Revised Child Anxiety and Depression Scale will be used. The raw score from the subscale, which ranges from 0-18, will be used to calculate the T score by taking into consideration development level and gender. A T score of 65 or higher indicates a score borderline the clinical threshold and a T score of 70 or higher indicates a score above the clinical threshold.

CONTACTS AND LOCATIONS:
Overall Officials: Lena J Xiao, MD, MSc, Principal Investigator — Provincial Health Services Authority British Columbia
Locations (1):
- British Columbia Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No